CLINICAL TRIAL: NCT02156635
Title: A Double-blind, Sham-controlled, Randomized Clinical Trial on Stroke Treatment Using Transcranial Direct Current Stimulation
Brief Title: Stroke Treatment Associate to Rehabilitation Therapy and Transcranial DC Stimulation
Acronym: START-tDCS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, MSc, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDCS 001
Record Dates: First submitted 2014-05-26; First posted 2014-06-05 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Stroke; Cerebrovascular Disorders; Cerebral Infarction
Keywords: Rehabilitation; Direct Current Stimulation; Acute Stroke
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Cerebral Infarction | interventions — Transcranial Direct Current Stimulation; Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tdcs / CIMT (Experimental): Participants in the acute post-stroke stage will receive active tDCS associate to rehabilitation (CIMT)
  Interventions: Device: Transcranial direct current stimulation; Behavioral: Constraint-Induced Movement Therapy
- Sham stimulation / CIMT (Sham Comparator): Participants in the acute post-stroke stage will receive sham stimulation associate to rehabilitation (CIMT)
  Interventions: Behavioral: Constraint-Induced Movement Therapy; Other: Placebo

INTERVENTIONS:
Device: Transcranial direct current stimulation
  Arms: Active tdcs / CIMT
Behavioral: Constraint-Induced Movement Therapy
Other: Placebo
  Arms: Sham stimulation / CIMT

SUMMARY:
The purpose of this study is to determine whether active stimulation of the affected hemisphere will be more effective than simulated current in treatment of stroke

DETAILED DESCRIPTION:
Stroke is defined as an acute neurological dysfunction of vascular origin, with subtle development of clinical signs of cerebral function disturbs, lasting more than 24h. The traditional therapy includes drugs and physical rehabilitation, without systematization, with complicates its replication. The transcranial direct current (DC) stimulation might promote an increase in the motor function of the hands, when compared with placebo stimulation.

In fact, some clinical trials point positive effects of transcranial DC stimulation (tDCS) as a post-stroke intervention, however, in general, they only include patients in the chronic stage, with cerebral damage in different areas and diverse disabilities, most being assisted by non-standardized physical therapy treatments. tDCS combined with a standardized physiotherapy program, noted as constraint-induced movement therapy (CIMT), could be able to modulate the cortical excitability and promote better functional recovery.

However, no relate of longitudinal studies assessing patients in the acute stage submitted to tDCS and physiotherapy for more than 6 months have been found. Studies like this would help us elucidate the action mechanisms of this treatment in the early stages of stroke.

With this in mind, START - tDCS, a phase II/III clinical trial, will be developed to assess the therapeutic effects of the tDCS in early stage enrolling 40 post-stroke patients. They will be allocated in 2 groups at random to receive active tDCS or sham, associate to CIMT. The protocol will be applied in a daily basis for 10 consecutive working days (2 weeks), after that, the patients will be followed for 1 month. By the end of the study, the participants that receive tDCS and show better clinical condition will be invited to participate in bimonthly stimulation for 12 months, as part of a longitudinal study regarding tDCS for stroke. An increase in the clinical condition will be considered as a final score higher than 10 points in the Barthel Index, our primary outcome, when compared with baseline, before the treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Ischaemic acute stroke
* Informed consent

Exclusion Criteria:

* 25 ≤ National Institute of Health Stroke Scale ≤ 32
* Rankim ≥ 5
* Mini Mental State Examination ≤ 24
* tDCS criteria: use of modulators of the Central Nervous System drugs; patients with implanted metallic or electronic devices; pacemaker; seizures; pregnancy;any other condition that might limit or interfere in the sensorimotor system CIMT criteria: inability to actively execute the movements of wrist flexion, metacarpophalangeal and interphalangeal active extension of 10º and wrist extension of 20º

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Functional Independence measured by Barthel Index | Change for functional independence at 4 months

SECONDARY OUTCOMES:
Cognitive dysfunction (Montreal Cognitive Assessment) | Baseline (week 1) and Endpoint (week 4)
Executive functions (Victoria version of the Stroop Color and Word Test) | Baseline (week 1) and Endpoint (week 4)
Attention and Working Memory (Digit span subtest) | Baseline (week 1) and Endpoint (week 4)
Spasticity | Baseline, Week 2 and Week 4
Muscle strength | Baseline, Week 2 and Week 4
Balance | Baseline, Week 2 and Week 4
Posture | Baseline, Week 2 and Week 4
Fear of falling during daily life activities | Baseline, Week 2 and Week 4
Upper limb function | Baseline, Week 2 and Week 4
Quality of life | Baseline, Week 2 and Week 4
Lower limb function | Baseline, Week 2 and Week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Paraíba,Department of Psychology, João Pessoa, Paraíba, Brazil

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411
- [Derived] Andrade SM, Santos NA, Fernandez-Calvo B, Boggio PS, Oliveira EA, Ferreira JJ, Sobreira A, Morgan F, Medeiros G, Cavalcanti GS, Gadelha ID, Duarte J, Marrocos J, Silva MA, Rufino T, Nobrega SR. Stroke Treatment Associated with Rehabilitation Therapy and Transcranial DC Stimulation (START-tDCS): a study protocol for a randomized controlled trial. Trials. 2016 Jan 28;17:56. doi: 10.1186/s13063-016-1186-7. PMID 26822418